CLINICAL TRIAL: NCT01810653
Title: A Double-blind, Randomized, Uninational, Multicenter, Two Parallel Groups, Active Controlled Study to Compare the Effect of the Treatment With Transipeg 2.95 g or Forlax Junior 4 g in Children With Constipation
Brief Title: A Study to Compare the Effect of Transipeg 2.95 g or Forlax Junior 4 g in Children With Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12052; 2015-000081-63 (EudraCT Number)
Record Dates: First submitted 2013-03-12; First posted 2013-03-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Constipation
Keywords: Macrogol
MeSH Terms: conditions — Constipation | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macrogol (Transipeg) (Experimental)
  Interventions: Drug: Macrogol (Transipeg, BAY81-8430)
- Macrogol (Forlax) (Active Comparator)
  Interventions: Drug: Macrogol (Forlax)

INTERVENTIONS:
Drug: Macrogol (Transipeg, BAY81-8430) — Up to 4 sachets per day based on individual titration
  Arms: Macrogol (Transipeg)
Drug: Macrogol (Forlax) — Up to 4 sachets per day based on individual titration
  Arms: Macrogol (Forlax)

SUMMARY:
The study design combines a long-term safety and a dose range determination objective. The first 8 weeks of the study were primarily intended for the dose range determination, while the later visits were used for the comparison of long-term safety between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Childhood functional constipation
* 6 months to <16 years of age
* Male or female
* For females of childbearing potential (after menarche): negative pregnancy test
* Moderately severe to severe constipation, defined as stool frequency <3 stools/week
* Informed consent signed by parent(s) or legal acceptable representative(s), after sufficient oral and written information before entering the study, to be documented by the investigators in the Case Report Form

Exclusion Criteria:

* Functional non-retentive fecal incontinence
* Known metabolic or endocrine disorders (s.a. hypothyroidism)
* Neurologic disorders (s.a. spina bifida or spinal cord anomaly)
* Hirschsprung's disease (congenital megacolon)
* Anal anomaly
* Gastrointestinal surgery
* Drug induced constipation
* Mental retardation
* Cerebral palsy
* Treatment with other laxatives
* Drugs influencing gastrointestinal function (e.g., cisapride, erythromicin, imodium)
* Prior bowel surgery, except appendectomy
* Earlier participation in this trial
* Concurrent participation in any other clinical trial
* Participation in any other clinical study 6 months prior to inclusion
* Any use of a Macrogol within 2 months prior to inclusion

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Symptom Based Weekly Total Sum Score (TSS) Over 52 Weeks | Baseline (Week 0), Week 1, 2, 3, 4, 8, 12, 26, 52
Change From Baseline in Total Sum Score (TSS) at Week 52 | Baseline, Week 52
Short Term Change of Total Sum Score (TSS): Average of Weeks 1 to 8 Minus Baseline | Average of Weeks 1 to 8
Long Term Change of Total Sum Score (TSS): Average of Weeks 26 and 52 Minus Baseline | Average of Weeks 26 and 52
Overall Change of Total Sum Score (TSS): Average of all Diaries Obtained Minus Baseline | Average up to 52 weeks
Dose Range Determination: Mean Dose Based on Sachets Used | Up to 52 weeks.
Dose Range Determination: Mean Dose per Kilogram Body Weight Based on Sachets Used | Up to 52 weeks

SECONDARY OUTCOMES:
Percentage of Treatment Success | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Defecation Frequency | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Consistency of the Feces | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Strains During Defecation | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Quantity of Stools | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Percentage of Subjects With Pain During Defecation | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Frequency of Pain (Times per Week) | Week 1, 2, 4, 8, 12, 26, 52
Percentage of Subjects With Abdominal Pain | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Frequency of Abdominal Pain (Times per Week) | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Relation of Abdominal Pain With Defecation | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Fecal Incontinence (Times per Week) and Fecal Incontinence (Times per Week) at Night | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Percentage of Subjects with Fecal Incontinence at Specified Time points | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Percentage of Subjects With Urgency for Defecation | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Frequency of Urgency for Defecation (Times per Week) | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Percentage of Subjects With Urine Incontinence (UI) During Day and Night | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Frequency of Urine Incontinence During Day and Night (Times per Week) | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Percentage of Subjects With Good, Moderate or Bad Appetite | Week 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Average Score for Diary Reported Diarrhoea | Week 0, 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Average Score for Diary Reported Flatulence | Week 0, 1, 2, 4, 8, 12, 26, 52
Individual Symptoms: Average Score for Diary Reported Nausea | Week 0, 1, 2, 4, 8, 12, 26, 52

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Netherlands (4):
  - Amsterdam
  - Eindhoven
  - Veldhoven
  - Woerden

REFERENCES:
- [Derived] Bekkali NLH, Hoekman DR, Liem O, Bongers MEJ, van Wijk MP, Zegers B, Pelleboer RA, Verwijs W, Koot BGP, Voropaiev M, Benninga MA. Polyethylene Glycol 3350 With Electrolytes Versus Polyethylene Glycol 4000 for Constipation: A Randomized, Controlled Trial. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):10-15. doi: 10.1097/MPG.0000000000001726. PMID 28906317
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/